CLINICAL TRIAL: NCT06567249
Title: Selective Intracoronary Hypothermia as a Prevention of Reperfusion Injury in ST-elevation Myocardial Infarction.
Brief Title: Intracoronary Hypothermia as a Prevention of Reperfusion Injury in Myocardial Infarction.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRI-262
Record Dates: First submitted 2024-08-18; First posted 2024-08-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction; ST-Elevation Myocardial Infarction (STEMI); Reperfusion Injury; Microvascular Occlusion
Keywords: hypothermia; ST-elevation myocardial infarction; microvascular obstruction; reperfusion injury; STEMI
MeSH Terms: conditions — Myocardial Infarction; ST Elevation Myocardial Infarction; Reperfusion Injury; Hypothermia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intracoronary hypothermia (Experimental): Selective intracoronary hypothermia starts by advancing the coronary guidewire beyond the occlusion of the culprit coronary vessel with subsequent over-the-wire balloon inflation at 5 atm at the site of the occlusion. Then, the guidewire is removed, and the infusion pump is connected to the over-the-wire balloon. Normal saline infusion starts with an infusion rate of 5 ml per minute and a duration of 5 minutes. The temperature of the saline is 4 °C. After that, the over-the-wire balloon is deflated, and infusion continues for 15 minutes at the same temperature and infusion rate of 5 mL per minute, followed by the standard percutaneous coronary intervention.
  Interventions: Procedure: Intracoronary hypothermia
- Conventional percutaneous coronary intervention (Other): The group will receive standard percutaneous coronary intervention.
  Interventions: Other: Standard percutaneous coronary intervention

INTERVENTIONS:
Procedure: Intracoronary hypothermia — This trial stands apart from other studies of intracoronary hypothermia, mainly because it will establish the role of intracoronary hypothermia in reducing infarct size not only in the left anterior descending artery territory but in other vessels as well, including the right coronary artery and circumflex coronary artery.
  Arms: Intracoronary hypothermia
Other: Standard percutaneous coronary intervention — Percutaneous coronary intervention is performed in a standard manner.
  Arms: Conventional percutaneous coronary intervention

SUMMARY:
Acute myocardial infarction with ST segment elevation is often accompanied by a totally occluded coronary artery. Which has deleterious effects on heart muscle. Primary percutaneous coronary intervention is the most effective mode of treatment for ST-elevation myocardial infarction (STEMI) patients. Despite the restoration of the blood flow, 30-60% of patients develop microvascular obstruction, which lowers the effects of the coronary blood flow restoration. The most advanced coronary microvascular obstruction presents as a no-reflow phenomenon, which is an abrupt deceleration or absence of coronary flow following stent implantation. Several pharmacological treatments have been proposed, as well as deferred stenting, but none of them really helped. Thus, new ways of alleviating coronary obstruction are warranted. One of the new ways of mitigating the reperfusion injury is intracoronary hypothermia, which showed to be safe on a handful of patients in small series. In the animal studies, intracoronary hypothermia demonstrated a protective effect in terms of reducing infarct area. But clinical studies failed to reproduce the protective effects of intracoronary hypothermia. Thus, our study, using a modified hypothermia protocol, will test the hypothermia hypothesis.

DETAILED DESCRIPTION:
The study aims to find the most effective methods for the prevention and treatment of microvascular obstruction and reperfusion injury, studying the pathophysiological mechanisms of the development of this complication is of key importance. Many of these mechanisms are now known. In particular, the risk of developing microvascular obstruction is directly proportional to the duration of coronary artery occlusion, the degree of platelet aggregation activity, and blood viscosity and is higher in patients with massive thrombosis of the ischemic artery during percutaneous coronary intervention, which suggests a significant contribution to the development of microembolization during mechanical thrombus fragmentation. Despite all the collected data, there is no effective mode of reperfusion injury prophylaxis. Thus, it is necessary to explore new ways of minimizing reperfusion injury during primary percutaneous coronary intervention. The goal of our study is to determine the safety and effectiveness of intracoronary hypothermia. All patients who meet the eligibility criteria for this study will be randomized in a 1:1 ratio to receive intracoronary hypothermia with subsequent percutaneous coronary intervention or a standard revascularization strategy. The total number of patients planned to be recruited is 60. The study was approved by the local ethics committee. The intracoronary hypothermia group will receive 4°C normal saline with an infusion rate of 5 ml/min for 5 minutes through the inflated over-the-wire balloon, followed by an infusion of 4°C normal saline for 15 minutes with the same infusion rate of 5 ml per minute through the deflated over-the-wire balloon. After that, standard percutaneous coronary intervention is performed. The control group will receive only the standard percutaneous coronary intervention procedure.

ELIGIBILITY:
Inclusion Criteria:

* Acute ST-elevation myocardial infarction
* Time from onset of symptoms less than 12 hours
* Given informed consent

Exclusion Criteria:

* Contraindication to MRI
* Cardiogenic shock
* Conduction disturbance: Atrioventricular block: 2nd and 3rd degree. SA block.
* Sick sinus syndrome requiring implantable pacemaker
* Pulmonary edema
* Active inflammatory condition
* Active chemo/radiation therapy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Infarct size (percent) | 7 days
  The primary endpoint is the infarct size, expressed as a percentage of total myocardium mass, revealed by the cardiac magnetic resonance imaging with late gadolinium enhancement after seven days.
Myocardial hemorrhage (percent) | 7 days
  Myocardial hemorrhage extent is visualized by T2-weighted sequences on cardiac magnetic resonance imaging and expressed as a percentage of total myocardium mass.
Microvascular obstruction (percent) | 7 days
  Microvascular obstruction is expressed as a percentage of total myocardium mass revealed by the cardiac magnetic resonance imaging with late gadolinium enhancement at day seven.

SECONDARY OUTCOMES:
Ejection fraction (percent) | 10 days
  Ejection fraction is measured by echocardiography and expressed as a percentage (Simpson's method).
Wall motion score index (score) | 10 days
  Wall motion score index (score) measured by echocardiography at day 10.

OTHER OUTCOMES:
Thrombolysis in myocardial infarction flow (score) | 1 hour
  Thrombolysis in myocardial infarction flow (score) assessed at the end of the primary coronary intervention on the scale from 0 to III.
Major adverse cardiac events (percent) | 30 days
  Incidence of major adverse cardiac events is expressed as a percentage.
Peak value of high-sensitivity troponin T (ng/L) | 5 days
  Peak value of high-sensitivity troponin T (ng/L) is measured in blood sample at day 5.
Conduction abnormalities (percent) | 5 days
  Total incidence rate of 2nd and 3rd degree atrioventricular block and sinoatrial block is expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Nasekina, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center; Vyacheslav Ryabov, Study Director — Cardiology Research Institute, Tomsk National Research Medical Center; Evgenyi Vyshlov, Study Chair — Cardiology Research Institute, Tomsk National Research Medical Center
Locations (1):
- Cardiology Research Institute, Tomsk National Research Medical Center, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.